CLINICAL TRIAL: NCT07213830
Title: An Open-label, Phase I/II First in Human, Dose Escalation, Optimisation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Anti-tumour Activity of IPN01203 in Participants With Locally Advanced or Metastatic Solid Tumours Who Have Progressed on or After Immune Checkpoint Inhibitor Therapies
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, Immunogenicity and Anti-tumour Activity of IPN01203 in Adults With Locally Advanced or Metastatic Solid Tumours Exposed to Immune Checkpoint Inhibitor Therapies
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CLIN-01203-450
Record Dates: First submitted 2025-10-01; First posted 2025-10-09 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: Part 1a is sequential assignment - non-randomized, single arm. Part 1b is randomized, two-arm, parallel design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase Ia: Dose Escalation (Experimental): Participants will receive assigned dose level IPN01203 administered intravenously (IV).
  Interventions: Biological: IPN01203
- Phase Ib: Dose Optimisation (Experimental): Participants will randomly receive one of the two doses of interest, determined at the end of Phase Ia, of IPN01203 administered intravenously (IV).
  Interventions: Biological: IPN01203

INTERVENTIONS:
Biological: IPN01203 — Study intervention will be provided in a vial.

SUMMARY:
The purpose of this study is to determine the appropriate dosage, safety and effectiveness of a new drug, IPN01203, in adults with advanced solid tumours.

Advanced solid tumours are cancers that can occur in various organs or tissues and have spread from their original site to nearby tissues or other parts of the body.

There will be two parts to this study:

* Phase Ia: This part (called dose escalation) will find the dose range that shows activity against the tumour and can be tolerated by participants by testing different increasing doses of IPN01203.
* Phase Ib: This part (called dose optimisation) will assess the ability of the drug to prevent, slow down, or stop the growth of tumours and how the body processes and responds to the drug when given in "low dose" or "high dose." It will also further explore the safety and tolerability.

An additional part (phase II) may be added to the study based on the results of phase Ia and phase Ib.

Each part will consist of the following periods:

* A screening period (up to 28 days) to assess whether the participant can take part, requiring at least 1 visit to the study centre.
* A treatment period where all eligible participants will receive IPN01203. Requires approximately 15 visits for the first 2 months followed by 3 visits every month from month 3 until unacceptable toxicity, disease progression, death, upon participant's withdrawal of consent, investigator decision, or study termination by the sponsor, whichever occurs first.

There will also be one visit at the end of treatment (EoT), 30 days after the last administration of the study intervention or prior to the start of new anticancer treatment, whichever is earlier. Additionally, there will be one visit (the safety follow-up visit) 90 days after the last administration of study intervention or prior to the start of new anticancer treatment, whichever is earlier.

In both parts of the study, participants will undergo blood sampling, urine collection, physical examinations and clinical evaluations. They may continue some other medications, but the details need to be recorded.

Each participant will be in this study until death or withdrawal from the study. IPN01203 will be provided to participants who tolerate it for as long as their disease does not progress. Participants may withdraw consent to participate at any time.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age, at the time of signing the informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Measurable disease per RECIST version 1.1 (at least one lesion that is measurable by RECIST 1.1. Tumour lesions in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions after radiation) and documented locally advanced or metastatic disease with CT and/or MRI.
* All acute, clinically significant (CS) treatment-related AEs from a prior therapy resolved to Grade 1 or lower prior to study entry. Participants with chronic toxicities such as Grade ≤2 neuropathy or alopecia can be included.
* Have a life expectancy for disease-related mortality, as evaluated by the investigator.
* Male and female participants: Contraceptive use by men or women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.
* Adequate haematologic and end organ function
* Participant is capable of giving signed informed consent as described in the protocol.

Exclusion Criteria:

* Have untreated or active primary brain tumour, Central Nervous System (CNS) metastases, leptomeningeal disease, or spinal cord compression.
* Experienced severe, life-threatening immune-mediated AEs, or infusion-related reactions such as those that lead to permanent discontinuation while on treatment with prior anticancer therapy such as immune checkpoint inhibitor therapy.
* History of known autoimmune disease
* History of stroke or significant cerebrovascular disease, encephalitis, meningitis, organic brain disease (e,g., Parkinson's disease) or uncontrolled seizures in the year prior to first dose of study drug.
* History of CS cardiac disease within 6 months prior to the initiation of study intervention, including but not limited to unstable angina, acute myocardial infarction, endoscopic or open-heart cardiac surgery, or heart failure classified as New York Heart Association Grade 2 or higher. Additional exclusion criteria include:

  1. Left ventricular ejection fraction <45%
  2. QT interval corrected by Fridericia (QTcF) >470 ms (for women) and >450 ms (for men) or CS arrhythmias.
* History of CS respiratory disease within 6 months prior to the initiation of study intervention, including severe chronic obstructive pulmonary disease or asthma.
* Prior organ transplantation.
* Chronic or ongoing active infections within 4 weeks prior to Cycle1 Day1 (C1D1).
* Presence of hepatitis B surface antigen (HBsAg) [or hepatitis B core antibody (HBcAb)] at screening or within 3 months prior to the first dose of study intervention.
* Positive hepatitis C antibody test result at screening or within 3 months prior to the first dose of study intervention.
* Participants with known history of HIV infection are excluded from the study unless they meet the following criteria:

  1. Stable Antiretroviral Therapy: Participants must be on a stable antiretroviral therapy regimen for at least 4 weeks prior to enrolment.
  2. CD4+ T cell Count: Participants must have a CD4+ T cell count of at least 200 cells/µL.
  3. Viral Load: Participants must have an undetectable viral load (HIV RNA <50 copies/mL)
  4. No Opportunistic Infections: Participants must not have had any opportunistic infections or other human immunodeficiency virus (HIV)-related illness within the past 6 months Note: HIV testing will be performed in any countries where it is mandatory per local requirements.
* History of other malignancy within the last years.
* Significant concurrent, uncontrolled medical condition that would put participants at unacceptable risk from study participation or preclude them from complying with study procedures per investigator including, but not limited to renal, hepatic, haematologic, gastrointestinal, endocrine, pulmonary, neurological, cerebral, or psychiatric disease.
* Treatment with >10 mg per day of prednisone (or equivalent) or other immune suppressive drugs within 7 days prior to the initiation of study drug. Exceptions may be made for participants who have had allergic reaction to iodinated contrast media. Steroids for topical, ophthalmic, inhaled, or nasal administration are allowed.
* Concurrent participation in another therapeutic treatment study.
* Participants accommodated in an institution because of regulatory or legal order; prisoners or participants who are legally institutionalised.
* For French participants only: participants are under court protection, not affiliated to a social security system or protected adults.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2032-07-14 (Estimated); Study Completion 2032-07-14 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with dose limiting toxicity (DLT) | Within 28 days of first dose
Percentage of participants experiencing treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TE-SAEs). | From the first IPN01203 administration to 90 days after the last dose.
  An Adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAE is an AE for which the start date is on or after the date that the intervention began
Phase Ib: Objective Response Rate (ORR) | At end of study (up to approximately 3 years)
  Defined as the percentage of participants with best overall response (BOR) of complete response (CR) or paritial response (PR), as determined by investigator per RECIST version 1.1.

SECONDARY OUTCOMES:
Phase Ia: Time to maximum observed drug concentration (Tmax) after single and multiple doses of IPN01203. | Up to 28 days after study drug administration.
Phase Ia: Maximum observed drug concentration (Cmax) after single and multiple doses of IPN01203 | Up to 28 days after study drug administration.
Phase Ia: Area under the plasma concentration time curve (AUCtau) after single and multiple doses of IPN01203. | Up to 28 days after study drug administration.
Phase Ia: Percentage of Treatment-Emergent Anti-Drug Antibodies (TEADA), Including Binding and Neutralizing Antibodies. | From the first dose of study drug administration, at predefined intervals until the end of study (up to approximately 3 years)
Phase Ia: Objective response rate (ORR) | At end of study (up to approximately 3 years)
  ORR is defined as the percentage of participants with BOR of CR or PR, as determined by investigator per RECIST version 1.1.
Phase Ib: Duration of response (DoR) | At end of study (up to approximately 3 years)
  DoR is defined as the time from first documented evidence of CR or PR until progressive disease, as determined by investigator per RECIST version 1.1, or death from any cause, whichever occurs first.
Phase Ib: Duration of stable disease (SD) | At end of study (up to approximately 3 years)
  SD is defined as the time from the date of first IPN01203 administration to the date of the first documented disease progression, as determined by investigator per RECIST version 1.1, or death due to any cause, whichever occurs first, for participants with SD as best response, with a minimum SD duration of 8 weeks.
Phase Ib: Progression-free survival (PFS) | At end of study (up to approximately 3 years)
  PFS is defined as the time from the date of first IPN01203 administration to the date of the first documented disease progression, as determined by investigator per RECIST version 1.1, or death due to any cause, whichever occurs first.
Phase Ib: Disease control rate (DCR) | From the first IPN01203 administration throughout the study (up to approximately 3 years).
  DCR is defined as the percentage of participants with BOR of CR, PR, or SD, as determined by investigator per RECIST version 1.1, from the first IPN01203 administration throughout the study.
Phase Ib: Time to response (TTR) | From the first IPN01203 administration throughout the study (up to approximately 3 years).
  TTR is defined as the time between date of start of treatment until first documented response (CR or PR), as determined by investigator per RECIST version 1.1.
Phase Ib: Percentage of Treatment-Emergent Anti-Drug Antibodies (TEADA), Including Binding and Neutralizing Antibodies. | From predose to end of treatment (up to approximately 3 years).

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (10):
- United States (5):
  - START MidWest PI Sharma, Grand Rapids, Michigan
  - Sarah Cannon Research Institute PI McKean Nasville, TN, USA, Nashville, Tennessee
  - MD Anderson PI Champiat, Houston, Texas
  - Start San Antonio PI Rasco, San Antonio, Texas
  - NEXT PI Spira, Fairfax, Virginia
- Princess Margaret Cancer Center PI Spreafico, Toronto, Canada
- Gustave Roussy Cancer Campus Grand Paris- (Institut de Cancerologie Gustave-Roussy) - PI Ronan, Villejuif, France
- Spain (3):
  - Hospital Universitario Vall d'Hebron PI Garralda Cabanas, Barcelona
  - NEXT Quiron-Barcelona - PI Saavedra Santa Gadea, Barcelona
  - START Madrid - CIOCC. Grupo Hospital de Madrid (HM) - Centro Integral Oncologico Clara Campal (CIOCC) - Calvo Aller, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, annotated case report form, statistical analysis plan, and dataset specifications.
  Patient level data will be anonymized and study documents will be redacted to protect the privacy of study participants.
Time Frame: Where applicable, data from eligible studies are available 6 months after the studied medicine and indication have been approved in the US and/or EU.
Access Criteria: Further details on Ipsen's sharing criteria and process for sharing are available here (https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/).
URL: https://www.ipsen.com/science/clinical-trials/clinical-data-transparency/